CLINICAL TRIAL: NCT06074926
Title: Promoting Healthier Food Acceptance and Intake Among Young Children Using a Novel Positive Parent-Child Interaction Strategy
Brief Title: Promoting Food Acceptance Through Positive Parenting: the Play and Grow Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Stephanie Anzman-Frasca, Associate Professor of Pediatrics, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007145
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Obesity, Childhood; Overweight, Childhood; Overnutrition; Pediatric Obesity; Eating, Healthy
Keywords: Repeated Exposure; Associative Conditioning; Positive Parenting; Food Acceptance; Diet Quality
MeSH Terms: conditions — Pediatric Obesity; Overnutrition

STUDY DESIGN:
Masking Description: Membership in the "intervention" versus "control" group will not be discussed as such, but participants will know whether they receive the repeated exposure (control group) or associative conditioning (intervention group) activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Intervention (Experimental): Participants will attend two laboratory visits and complete a 3-week intervention, which consists of interactive parent-child activities (~45 min of interactive activities/week) that pair tasting an assigned target vegetable with positive parent-child interactions. Positive interactions will be promoted via positive parenting prompts embedded in the activity instructions (e.g., prompts promoting child-directed play).
  Interventions: Behavioral: Associative Conditioning
- Group 2 - Control (Experimental): Participants will attend the same two laboratory visits and complete a 3-week intervention, which consists of only individual taste exposures to their target vegetable.
  Interventions: Behavioral: Repeated Exposure

INTERVENTIONS:
Behavioral: Associative Conditioning — There will be 3 planned activities per week (9 total) within play kits provided to families. Children will first taste their assigned target vegetable and then complete an activity with their parent following provided instructions. Activity instructions will include positive parenting skills adapted from evidence-based parenting programs (i.e., Parent-Child Interaction Therapy (PCIT) and Triple-P) designed to promote positive parent-child interactions.
  Arms: Group 1 - Intervention
Behavioral: Repeated Exposure — There will be 3 planned exposures per week (9 total). Exposures will include only individual tastes of the child's assigned target vegetable.
  Arms: Group 2 - Control

SUMMARY:
Approximately one half of adults and one-fifth of children have obesity, including 14% of 2-5-year-olds. Early obesity prevention is essential as children who are overweight by age 5 are at increased risk for later obesity. Dietary intake is inextricably linked to weight status, and the majority of young children fail to meet intake recommendations, with socioeconomically disadvantaged and racial/ethnic minority children at increased risk of poor diet quality. However, children's liking of healthier foods predicts their intake, and children can learn to like healthier foods via experience. The current study brings together evidence from the parenting and learning literatures to: 1) examine effects of a novel learning strategy leveraging positive parent-child interactions on 3-5-year-old children's vegetable acceptance and dietary intake, as well as to explore 2) individual differences in learning strategy effects.

DETAILED DESCRIPTION:
Repeated exposure, in which children taste a target food across several occasions, is an effective strategy for increasing children's acceptance and intake of healthier foods. An alternative strategy that may be preferable for those less likely to try unfamiliar or disliked foods is associative conditioning. This refers to changes in one's response to a target food after it is repeatedly, concurrently paired with an unconditioned stimulus - typically another food - that already has a positive valence. While evidence-based, this approach has the disadvantage of adding extra calories and exposure to less healthy foods.

Pilot data provided support for the hypothesis that non-food stimuli could be leveraged in conditioning strategies to promote healthier food acceptance. After pairing positive peer interactions (via group games) with tasting a target vegetable across 11 sessions, 6-8-year-old children's preferences for target vegetables increased at post-test. In considering application of this approach for younger children, positive parent-child interactions may be an appropriate non-food stimulus as parents are a primary social influence for this age group. Despite this, no studies to date have leveraged this positive stimulus in the context of associative conditioning paradigms designed to promote vegetable acceptance. Additionally, although other food preference learning approaches, like repeated exposure, are well-established in the experimental literature, less is known regarding individual differences impacting intervention effectiveness.

The current study seeks to examine effects of a novel learning strategy leveraging positive parent-child interactions on 3-5-year-old children's vegetable acceptance and dietary intake, as well as to explore individual differences in learning strategy effects. Findings will inform future intervention work, as well as offer insight into potential behavioral factors influencing young children's diet and health.

ELIGIBILITY:
Inclusion Criteria:

* Child is 3-5 years old
* Parent/ guardian is 18 years of age or older
* Child is not diagnosed with a serious physical or mental health condition that precludes safe participation
* Parent and child are English speaking

Exclusion Criteria:

* The child is outside the age range of 3-5 years
* Child is diagnosed with a serious physical or mental health condition that precludes participation
* Parent/ guardian is less than 18 years of age

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Child's target vegetable preference | Week 5 (post-test)
  Ranked ordered preference overall (range 1-7, 7 = least preferred) and relative to control vegetable
Child's target vegetable liking | Week 5 (post-test)
  Child-reported liking (3-point visual face scale (e.g., yummy, yucky, just OK) adapted from Birch and colleagues) overall and relative to control vegetable
Child's willingness to taste target vegetable | Week 5 (post-test)
  Observed by study staff, defined as child placing vegetable in his/her mouth (i.e., eating the vegetable or spitting it out)
Child target vegetable ad libitum consumption | Week 5 (post-test)
  10-minute period where child can eat as much or as little of provided foods (7 study vegetables + a neutral snack food (i.e., cracker)). Consumption will be measured via plate waste and overall consumption (grams) of the target vegetable, as well as consumption relative to the a) control vegetable and b) neutral snack will be calculated

SECONDARY OUTCOMES:
Reported general parenting | Week 5 (post-test)
  Parents will complete the Comprehensive General Parenting Questionnaire (CGPQ; items rated from 1 (strongly disagree) - 5 (strongly agree), higher scores reflect higher level of parenting dimension of interest) to assess 5 dimension of general parenting (sensitivity/nurturance, structure, overprotection, coercive control, behavioral control)
Observed general parenting | Week 5 (post-test)
  Observations of parenting will be coded from an 8-minute interactive play activity using the Iowa Family Interaction Rating Scales (IFIRS; ratings range from 1-9, 9=higher levels of behavior of interest). Aspects of parenting examined include: positive mood, warmth/support, physical affection, communication, listener responsiveness, prosocial behavior, encourages independence, intrusiveness, positive reinforcement, sensitive/child-centered, relationship quality
Observed child affect/behavior | Week 5 (post-test)
  Observations of child affect/behavior will be coded from an 8-minute interactive play activity with a parent using the IFIRS Scales (described previously). Aspects of child affect/behavior examined include: positive mood, prosocial behavior, antisocial (i.e., externalizing) behavior

OTHER OUTCOMES:
Frequency of vegetables consumed by child (past week) | Week 4 (intervention period)
  Parents will report on how often their child consumed vegetables during week 4 (intervention period) via the EPOCH Preschooler Dietary Questionnaire (range: 0 to "more than once per day")
Variety of vegetables consumed by child (past week) | Week 4 (intervention period)
  Parents will report which of 26 possible types of vegetables their child consumed during week 4 (intervention period) via the EPOCH Preschooler Dietary Questionnaire (range: 0 to 26)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Anzman-Frasca, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No